CLINICAL TRIAL: NCT03135236
Title: Parents as the Primary Sexuality Educators for Their Young Adults With Down Syndrome: The Effectiveness of a Family-based Training
Brief Title: Parents as the Primary Sexuality Educators for Their Young Adults With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AdvocateHC
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2018-06

CONDITIONS: Down Syndrome; Intellectual Disability; Sexuality; Parent-Child Relations
Keywords: Parent training; Family education; Young adults; Down syndrome; sexuality
MeSH Terms: conditions — Down Syndrome; Intellectual Disability; Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent training (Experimental): All registered participants will participate in a series of trainings (3 separate) on sexuality education.
  Interventions: Behavioral: Parent training

INTERVENTIONS:
Behavioral: Parent training — Participants will attend 3 trainings. There will be a pre-test before training 1 and an initial post-test after training 3. There will be a final post-test 1 month after the final training.

SUMMARY:
By integrating sexuality and disability literatures, theories, and research methodologies, this study aims to: 1) contribute to the limited knowledge professionals have of parents as the primary sexuality educators; 2) create a resource for parents in order to be sexuality educators for their young adults with I/DD; and 3) evaluate the effectiveness of the Home B.A.S.E. for Developmental Disabilities Curriculum.

In order to meet the objectives the study seeks to answer the following questions:

1. What is the effectiveness of a sexuality education workshop for parents of young adults with DS on improving the self-efficacy and attitudes around sexuality and healthy relationships for young adults with DS as well as increase the parent-child communication on sexuality topics?
2. What are parents' concerns that impact their ability to be the primary sexuality educators for their young adults with DS? It is proposed that parent confidence and comfort talking about sexuality topics with their young adult with Down syndrome will increase thereby increasing the parent-child communication as a result of this study.

DETAILED DESCRIPTION:
Enrollment will begin and will end once 30 eligible subjects have been identified. Anticipated duration is one year. Participants will enroll in one of the 4 different training series. Each series will have 3 dates they must attend. Once enrolled and consent is documented, eligible subject's will participate in the study for approximately three months. Participants will be expected to attend 3 training sessions over a 4 week period, each are up to 3 hours in length. There will be a follow-up post-survey one month after the last training and an optional phone interview that will occur 2 months after the final training. Participants will be compensated for their time with a $50 gift card once the final post-survey has been received. The gift card will be mailed to the family. Data analysis will begin once all trainings have been completed. Investigators anticipate completing the study, including primary analyses, within two years from the date recruitment begins.

ELIGIBILITY:
Inclusion Criteria:

* Parents of young adults with Down syndrome ages 20-30.
* Be able to communicate in English

Exclusion Criteria:

* Parents of young adults between the ages of 20 and 30 without Down syndrome
* Parents of individuals with Down syndrome younger than 20 or older than 30.
* Parents unable to attend 3 training sessions.
* Not fluent English communicators.
* Any vulnerable populations including pregnant women, neonates, prisoners, children, cognitively impaired adults, or adults unable to consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Pre-survey, post-survey, and final post-survey | 15-20 minutes
  A paper survey will be completed before training 1 that gathers quantitative data that will address attitudes, self-efficacy, and behaviors of the parents in attendance. The survey will also be completed at the end of training 3 and then mailed to the participant to complete 1 month after the final training. The quantitative data will be used to measure a change in the attendees' attitudes, confidence, and behaviors before and after the proposed intervention. Data will be analyzed using SPSS.

SECONDARY OUTCOMES:
Qualitative data | 5-15 minutes
  Qualitative data will be collected at the end of the first and second training session with two to three take home open-ended questions for each participant to answer as well as after the training is over with open ended questions on the initial follow-up survey. Structured phone interviews will be completed with a small sample of the participants after the one month follow-up paper survey. Answers and interview questions will be transcribed, coded, and themes will be established.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Frank, PhD, OTR/L, Principal Investigator — Advocate Healthcare
Locations (1):
- Advocate Adult Down Syndrome Center, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Bundy, M. L., White, P.N. (1990). Parents as sexuality educators: A parent training program. Journal of Counseling & Development, 68: 321-323.
- [Background] Frank, K. E. (2016). Parents as the primary sexuality educators for their adolescents with Down syndrome. (Doctoral dissertation). University of Illinois at Chicago, Chicago, IL. Retrieved from Indigo at http://hdl.handle.net/10027/21214.
- [Background] Klein JD, Sabaratnam P, Pazos B, Auerbach MM, Havens CG, Brach MJ. Evaluation of the parents as primary sexuality educators program. J Adolesc Health. 2005 Sep;37(3 Suppl):S94-9. doi: 10.1016/j.jadohealth.2005.05.004. PMID 16115575
- [Background] Raffaelli M, Bogenschneider K, Flood MF. Parent-teen communication about sexual topics. J Fam Issues. 1998 May;19(3):315-33. doi: 10.1177/019251398019003005. PMID 12295941